CLINICAL TRIAL: NCT05577871
Title: Echocardiographic Evaluation of the Effect of Dexmedetomidine Infusion as an Adjuvant to General Anesthesia in Off-pump Coronary Artery Bypass Grafting
Brief Title: Dexmedetomidine in Off Pump Coronary Artery Bypass Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dex in CABG
Record Dates: First submitted 2022-10-08; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dex group (Active Comparator): patients medicated with dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- control group (Placebo Comparator): patients took placebo normal saline.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — infusion of dexmedetomidine during the off pump coronary artery bypass grafting surgery
  Arms: dex group
Drug: normal saline — infusion of normal saline during the off pump coronary artery bypass grafting surgery
  Arms: control group

SUMMARY:
the study will assess the impact of intraoperative dexmedetomidine infusion on myocardial performance by investigating the left ventricular (LV) systolic and diastolic function and right ventricular (RV) fraction area change (which reflect RV systolic function) using two-dimensional trans-esophageal echocardiography (TEE) in patients undergoing elective first-time isolated off-pump coronary artery bypass (OPCAB) grafting. LV Systolic function will be measured by the TEE via the fractional area change, fraction shortening, and ejection fraction.

DETAILED DESCRIPTION:
Off pump coronary revascularization is an old technique performed first in St Petersburg in 1964, Off pump coronary artery surgery has been developed following two different approaches. Minimally invasive direct-access coronary artery bypass (MIDCAB) that consists of anastomosing the left internal mammary artery to the left anterior descending coronary artery through small anterior left thoracotomy, The second approach is multi-vessel grafting without CPB performed through standard median sternotomy. Dexmedetomidine (Dex), a highly selective α2-adrenergic receptor agonist, is widely used for sedation and analgesia in the ICU or as an anesthetic adjuvant.

This study will be a prospective comparative controlled randomized double blinded clinical trial on 36 patients divided into control ,and dexmedetomidine group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective first-time off-pump isolated coronary artery bypass graft (OPCAB) surgery
* Patients with good ventricular functions.
* Patients with normal levels of cardiac troponin I and myocardial enzymes
* Patients of Body Mass Index (BMI) more than 20 and less than 34.

Exclusion Criteria:

* Severe functional liver or kidney disease.
* Diagnosed HF (NYHA class >3).
* Arrhythmia or received treatment with anti-arrhythmic drugs.
* Severe bradycardia (HR < 45 bpm) and AV block.
* Pathologic esophageal lesion (esophageal stricture or varix )
* Pregnancy.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fraction | immediatly after sternal closure
  using transesophageal echocardiography, ejection fraction will be assessed by the ratio of stroke volume and end diastolic volume
left ventricular fractional shorting | immediatly after sternal closure
  using transesophageal echocardiography, fractional area change of the left ventricle will be calculated
left ventricular diastolic function | immediatly after sternal closure
  using transesophageal echocardiography, diastolic function (filling ratio) will be assessed by the ratio between early transmitral flow (E) and mitral annular tissue velocity (E').

SECONDARY OUTCOMES:
right ventricular systolic function | immediatly after sternal closure
  right ventricular systolic function assessed by (fraction area change) as assessed using transesophageal echocardiography.